CLINICAL TRIAL: NCT01851304
Title: Checking Melanoidins and Bitter Compound Satiating Efficiency Through Evaluation of Human Gut-brain Response to Novel-food Ingestion
Brief Title: Metabolic Effect of New Foods Through Gut-brain Axis
Acronym: CHECKMATE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Paola Vitaglione, Dr, Federico II University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: CKMPON-013
Record Dates: First submitted 2013-05-08; First posted 2013-05-10 (Estimated); Last update posted 2015-10-02 (Estimated); Status verified 2015-09

CONDITIONS: Obesity; Overweight
Keywords: beta-Glucans; Bitter; Bread; Coffee; Gentiana lutea; Melanoidins; Microencapsulation
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- Control Bread (Placebo Comparator): A 100 g portion of Control Bread with no extra fiber added. The control bread will be consumed in the intervention Satiety of breads
  Interventions: Dietary Supplement: Satiety of breads
- Bread Crust Bread (Experimental): A 100 g portion of Bread Crust Bread with 3 g bread crust per 100 g portion of control bread. The bread crust bread will be consumed in the intervention Satiety of breads.
  Interventions: Dietary Supplement: Satiety of breads
- Coffee Melanoidins Bread (Experimental): A 100 g portion of Coffee Melanoidins Bread with 3 g of isolated coffee melanoidins per 100 g portion of control bread. The coffee melanoidins bread will be consumed in the intervention Satiety of breads.
  Interventions: Dietary Supplement: Satiety of breads
- beta-Glucans Bread (Experimental): A 100 g portion of beta-Glucans Bread with 3 g of barley beta-glucans per 100 g portion of control bread. The beta-glucans bread will be consumed in the intervention Satiety of breads.
  Interventions: Dietary Supplement: Satiety of breads
- Control Pudding (Placebo Comparator): A 150 g portion of Control Pudding without the addition of any extracts. The control pudding will be consumed in the intervention Satiety of puddings.
  Interventions: Dietary Supplement: Satiety of puddings
- Gentian extract pudding (Experimental): A 150 g portion of Gentian Pudding with the addition of 1 g Gentian extract per 100 g pudding. The Gentian extract pudding will be consumed in the intervention Satiety of puddings.
  Interventions: Dietary Supplement: Satiety of puddings
- Encapsulated Gentian Extract Pudding (Experimental): A 150 g portion of Microencapsulated Gentian extract pudding with the addition of 1 g of a microencapsulated Gentian extract per 100 g pudding. The Microencapsulated Gentian extract pudding will be consumed in the intervention Satiety of puddings.
  Interventions: Dietary Supplement: Satiety of puddings

INTERVENTIONS:
Dietary Supplement: Satiety of breads — One separate breakfast session to consume each bread along with 125 mL skim milk. The session will start after an overnight fast followed by 5 separate blood draws over a 3 hour period before a provided lunch.
  Arms: Bread Crust Bread; Coffee Melanoidins Bread; Control Bread; beta-Glucans Bread
Dietary Supplement: Satiety of puddings — One separate breakfast session will be used to evaluate satiating efficacy of puddings after an overnight fast. After pudding consumption, five separate blood draws will be taken over a 3 hour period before a provided lunch.
  Arms: Control Pudding; Encapsulated Gentian Extract Pudding; Gentian extract pudding

SUMMARY:
A diet high in easily obtained energy-dense foods leads to the problems of overweight and obesity common in the developed world. Foods enriched with fiber or bitter compounds may increase satiety and decrease energy intake. This intervention will measure the effectiveness of coffee melanoidins, bread melanoidins, beta-glucans, and a Gentiana lutea L. extract in both a free or encapsulated form to decrease energy intake and modify the physiological markers of satiety in the short term. In particular bread (fiber) and a pudding (Gentiana lutea L. extract) will be used as tasty food matrices in the study.

DETAILED DESCRIPTION:
Overweight and obesity are health problems of utmost importance to the world population. The continuous development and consumption of high-energy foods at a low cost is correlated with an increased risk of diabetes and insulin resistance in addition to weight gain. To maintain body weight, a balance between energy intake and energy expenditure must be obtained. Since weight gain is a common outcome with an energy-dense diet, the best approach to reduce caloric intake is through the consumption of fruits and vegetables. However, this approach is usually unsatisfactory in the long-term as the loss of tasty food and the low reward of healthy meals often undermines the nutritionally prudent diet. A possible alternative approach is to produce tasty foods with low caloric density and satiety-inducing compounds that can reduce caloric intake and increase the sensation of satiety.

The human body regulates energy intake through a complex and interconnected biological system involving gut-brain axis, the endocannabinoid system and the hypothalamic-pituitary-adrenal axis. Biomarkers in the hypothalamic-pituitary-adrenal axis regulate food intake and the physiological response to stress. In the absence of food, the brain senses hunger through the elevation of the gastrointestinal hormone ghrelin. Once food is ingested, ghrelin levels decrease while other biomarkers in the gut-brain axis are released to increase feelings of satiety through the delay of gastric emptying, decrease in appetite and the decrease in food intake. Recent studies in mice have linked the endocannabinoid system with the hypothalamic-pituitary-adrenal axis through physiological stress and energy homeostasis. Furthermore, the endocannabinoids anandamide and 2-arachidonoylglycerol are both elevated during hunger but decrease after feeding.

Natural foods with low energy density, such as fruits and vegetables, usually contain a high amount of dietary fiber. Dietary fiber is classified as either soluble fiber (beta-glucans) or insoluble fiber (wheat bran) but both soluble and insoluble fiber have been strongly linked to increased satiety sensation. Dietary fiber is important for a properly functioning gastrointestinal tract by providing a nutrient source for bacteria in the large intestine. When a 3% portion of barley beta-glucans were added to a fruit drink or to bread and consumed at breakfast, a reduction in energy intake of 30% over 24 hours was observed along with beneficial changes in post-prandial gastrointestinal hormones involved in the biological control of hunger and satiety. Intake of insoluble fiber improves insulin sensitivity and enriched barley fiber bread or wheat fiber bread improved ghrelin and peptide YY (PYY) hormone response compared to control bread. A recently characterized class of food compounds, melanoidins, have been found to exhibit similar properties to dietary fiber in the gastrointestinal tract. Melanoidins are formed by the Maillard reaction process through the reaction of proteins with reduced carbohydrates and sugars during the cooking of heat-treated foods. Melanoidins are large insoluble or partially insoluble complexes that are present in coffee, bread, cocoa, and beer. However, the main sources of melanoidins in the diet are from coffee and bread with a contribution of 0.5-2.0 g/day of coffee melanoidins and 1.8-15 g/day of bread melanoidins. Research has shown that coffee melanoidins are fermented in the gastrointestinal tract while bread melanoidins stimulate bifidobacteria in the large intestine.

Bitter compounds have also been recently implicated in increasing satiety and having a beneficial effect on gastrointestinal tract hormones. Recent research in animals indicates that several bitter compounds can reduce the rate of gastric emptying, induce the secretion of satiety-inducing hormones cholecystokinin and glucagon-like peptide 1 (GLP-1), and decrease food intake. However, the animal experiments required the bitter compounds to be delivered directly to the stomach for action. A few bitter tasting vegetables, including broccoli and chicory, show beneficial health effects. Some natural phytochemicals are polyphenols known to possess different biological mechanisms and to have a bitter taste. The plant species Gentiana lutea L. produces several biologically active bitter phytochemicals, including the iridoid (loganic acid) and the secoiridoids (swertiamarin, gentiopicroside, amarogentin, sweroside). Gentiana lutea L. is used most often for the production of herbal teas and liqueurs.

In this randomized, crossover trial, the hunger and satiety feelings will be measured while blood will be collected at specific time points during the seven arms. Since this intervention is to develop tasty foods that both increase satiety and decrease energy intake in the short term, the bitter compounds will also be encapsulated in a protective coating. Encapsulation is commonly used to protect pharmaceuticals during passage through the oral cavity or stomach to enable the active compounds to be properly absorbed in the body. The coating used in one arm will allow the Gentiana lutea L. extract to pass through the oral cavity, allowing the volunteers to not taste the bitter compounds, for target in the stomach and duodenum.

All volunteers will participate in the seven arms of the study. Three different fiber-enriched breads and a control bread will be consumed in addition to skim milk at breakfast in four interventions. In the other three interventions, participants will consume a control pudding, Gentiana lutea L. extract pudding and the encapsulated Gentiana lutea L. extract pudding. A one-week washout period will be included between two separate interventions. The hedonic feelings of satiety, hunger, and appetite will be measured with a questionnaire at time 0 (baseline) and at 0.5, 1, 2, and 3 hours after breakfast. After 3 hours, the volunteers will consume lunch until they are satiated and then keep a food diary to record their intake throughout the rest of the day. In addition, blood will be collected at each time point and the amount of the specific hormones, neuropeptides, and endocannabinoids will be measured as part of the secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Normal body weight: Body Mass Index between 20 - 30
* Healthy by medical assessment
* Signed a written informed consent form
* Habitually consumes breakfast

Exclusion Criteria:

* Pregnant or breast feeding
* Diagnosed with intestinal or metabolic diseases/disorders, such as diabetes, renal, hepatic or pancreatic disorders, or ulcers
* Has hypertension or high cholesterol
* Food allergies and food intolerances including celiac disease and lactose intolerance
* Previous abdominal or gastrointestinal surgery
* Regular consumption of medication or drugs (including cannabis)
* Antibiotic or prebiotic therapy within the previous 2 months of the study
* Unwillingness to consume experimental foods
* Concurrent participation or previous participation in another clinical trial during the past year

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2014-09; Primary Completion 2015-07 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Variation in the feelings of appetite | 0, 0.5, 1, 2, and 3 hours
  Measure of the satiating effect for each bread and pudding with Visual Analog Scale (Area Under the Curve) over time for hunger, fullness and satiety.

SECONDARY OUTCOMES:
Variation in neuropeptide markers | 0, 0.5, 1, 2, 3 hours
  Measure serum beta-endorphin, neurotensin, orexin A, substance P, oxytocin, melatonin, alpha-melanocyte-stimulating hormone (pg/mL) and area under the curve (AUC) over time.
Variation in stress markers | 0, 0.5, 1, 2, 3 hours
  Measure serum cortisol (pg/mL) and area under the curve (AUC) over time.
Variation in serum endocannabinoids | 0, 0.5, 1, 2, 3 hours
  Measure serum anandamide, oleoylethanolamide, palmitoylethanolamide, linoleoyl ethanolamide (pg/mL) and area under the curve (AUC) over time.
Variation in salivary enzyme activity | 0, 0.5, 1, 2, 3 hours
  Measure salivary lipase (U/L) and salivary alpha-amylase (U/mL) activity.
Variation in salivary endocannabinoids | 0, 0.5, 1, 2, 3 hours
  Measure salivary anandamide, oleoylethanolamide, palmitoylethanolamide, linoleoyl ethanolamide (pg/mL)
Variation in gastrointestinal markers | 0, 0.5, 1, 2, 3 hours
  Measure serum ghrelin, peptide YY, glucagon-like peptide 1 (GLP-1), pancreatic polypeptide (PP), amylin, gastric inhibitory polypeptide (GIP), leptin, insulin (pg/mL)and area under the curve (AUC) over time.

CONTACTS AND LOCATIONS:
Overall Officials: Paola Vitaglione, Dr, Study Director — University of Naples
Locations (1):
- Department of Agriculture and Food Science, Portici, Italy